CLINICAL TRIAL: NCT07115420
Title: Optimising EUS-guided Choledochoduodenostomy With Lumen Apposing Metal Stent With Stent in Stent Placement: a Randomised Study Between Double Pigtail Stent and Fully Covered Self-Expanding Metal Stent. The Opti-LAMS Study
Brief Title: Improving a Bile Duct Drainage Procedure in Patients With Inoperable Cancer Blocking the Bile Ducts: Comparing Two Types of Endoscopically Placed Internal Stents to Prevent Blockage of a Lumen Apposing Metal Stent
Acronym: Opti-LAMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Waikato Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RD025065
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Malignant Biliary Obstruction; Advanced Pancreatic Cancer and Cholangiocarcinoma; Inoperable Malignant Biliary Obstruction; Lumen Apposing Metal Stents
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fully covered self expanding metal stent (FCSEMS) within LAMS (Experimental): In those randomised to FCSEMS, size will depend on the size of the LAMS with a 6mm LAMS to be stented with 8mm diameter FCSEMS and an 8mm LAMS to be stented with a 10mm FCSEMS, 4cm or 6cm length. The aim is to have at least 3cm of FCSEMS in the duodenal lumen If unable to place FCSEM through LAMS, crossover to DPS is allowed with plan for both intention to treat and per protocol analysis to be undertaken after completion of the study
  Interventions: Device: Fully covered self expanding metal stent (FCSEMS) within LAMS
- Double pigtail stent (DPS) within LAMS (Active Comparator): In those randomised to DPS, a double pigtail will be placed through the LAMS. The size of the stents will be left to the discretion of the proceduralist though 7Fr calibre with 7cm length is the recommended size
  Interventions: Device: Double pigtail stent (DPS) within LAMS

INTERVENTIONS:
Device: Fully covered self expanding metal stent (FCSEMS) within LAMS — In those randomised to FCSEMS, size will depend on the size of the LAMS with a 6mm LAMS to be stented with 8mm diameter FCSEMS and an 8mm LAMS to be stented with a 10mm FCSEMS, 4cm or 6cm length. The aim is to have at least 3cm of FCSEMS in the duodenal lumen If unable to place FCSEM through LAMS, crossover to DPS is allowed with plan for both intention to treat and per protocol analysis to be undertaken after completion of the study
  Arms: Fully covered self expanding metal stent (FCSEMS) within LAMS
Device: Double pigtail stent (DPS) within LAMS — In those randomised to DPS, a double pigtail will be placed through the LAMS. The size of the stents will be left to the discretion of the proceduralist though 7Fr calibre with 7cm length is the recommended size
  Arms: Double pigtail stent (DPS) within LAMS

SUMMARY:
This study looks at the best way to treat bile duct blockage in people with advanced cancer that cannot be removed by surgery. A blocked bile duct can cause serious symptoms like yellowing of the skin (jaundice), infection, and pain.

A common procedure called ERCP sometimes doesn't work in these patients. A newer method called EUS-guided choledochoduodenostomy (EUS-CDS) uses internal ultrasound to place a special metal tube (called a LAMS) to allow bile to drain. However, over time this stent can still become blocked.

To reduce this risk, doctors can place a second stent inside the first. This study is comparing two types of these second stents:

* A plastic stent (double pigtail stent or DPS)
* A metal stent (fully covered self-expanding metal stent or FCSEMS)

The study will include patients at Waikato Hospital. After the first stent is placed, they will be randomly assigned to receive either a DPS or FCSEMS. Patients will be followed for 6 months to see how well the stents work.

The aim is to find out which approach keeps the bile duct open longer and reduces the need for further procedures or hospitalisation, helping improve care and comfort for people with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Radiologically or histologically proven malignant distal bile duct obstruction with unresectable or metastatic disease, including those who have already failed ERCP
* Indication for biliary drainage with presence of obstructive jaundice biochemically and dilated biliary system on imaging.
* Informed consent provided.
* Common bile duct (CBD) size of at least 12mm on EUS imaging

Exclusion Criteria:

* Previous biliary stenting or surgery precluding EUS-CDS.
* Inability to provide informed consent.
* Pregnancy.
* Significant coagulopathy that is not correctable.
* Futility of intervention e.g. pre-terminal patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of stent dysfunction (defined as recurrent jaundice and/or cholangitis) in patients with malignant biliary obstruction receiving FCSEMS vs DPS stent-in-stent through LAMS | 26 weeks

SECONDARY OUTCOMES:
Technical success of LAMS placement. | 1 day
  Whether the LAMS stent is able to be successfully placed in the procedure
Technical success of second stent-in-stent placement | 1 day
  Whether the second stent (either FCSEMS or DPS) is able to be placed successfully
Clinical success of biliary drainage (evaluated at weeks 1, 2, 4, 12, and 26 using bilirubin and liver enzymes). | weeks 1, 2, 4, 12, and 26
  whether biliary drainage has been successful based on biochemical blood tests
Re-intervention rate | 26 weeks
  blockage of the LAMS stent requiring repeat procedure(s) as evidenced by clinical, biochemical evidence, and/or radiological evidence of biliary obstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Waikato Hospital, Te Whatu Ora Health New Zealand Waikato, Hamilton, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 3 months after time of publication for 5 years
Access Criteria: Other researchers will be able to access the above documents but no identifying patient data. They will have to email the head investigator to request the information, citing the reason for the request, and the head investigator will decide whether to grant access to the information or not